CLINICAL TRIAL: NCT06531031
Title: Clinical Performance Study of Microbio InfectID-BSI for Detection of Bacteria and Yeast
Brief Title: Clinical Performance Study of Microbio InfectID-BSI for Detection of Bacteria and Yeast With Patient Blood Samples
Acronym: IID-BSIqPCR
Status: Not yet recruiting | Type: Observational
Sponsor: Microbio Co Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MB-CLA-PRT-0022
Record Dates: First submitted 2024-07-24; First posted 2024-07-31 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Bloodstream Infection; Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — An additional 2 x EDTA tube will be collected at the same time as routine bloods are collected for suspected sepsis. One EDTA tube will be collected for the purposes of testing on the InfectID-BSI assay, and the 2nd EDTA tube will be collected for the purposes of storing the sample to aid in DNA sequencing for discordant results between InfectID-BSI and standard of care blood cultures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: InfectID-BSI (Bloodstream Infection) qPCR Assay — InfectID-BSI technology targets nucleic acid sequences unique to the target analyte. The qPCR raw data collected from InfectID-BSI's 9 assay tubes is analysed by Microbio's InfectID-Client (InfectID-BSI-associated software) and the result is reported as an analyte-detection if the unique target analyte is present or no result if the unique target analyte is absent.
  InfectID-BSI is carried out with whole blood from a venous puncture (EDTA). DNA is extracted from a sample of the collected blood using a validated DNA extraction instrument according to the manufacturer's instructions. The extracted DNA is then added to the InfectID-BSI qPCR reagent panel which consists of 9 reaction tubes (6 for bacteria, and 3 for yeast species). The panel is subjected to real-time qPCR using a process of Melt Curve analysis using the Rotor-Gene Q MDx qPCR instrument. The assay report identifies the species present in the sample upon completion. Results are generated within 3 hours.

SUMMARY:
The objective of the study is to determine the efficacy of the Microbio InfectID-BSI qPCR kit in a clinical laboratory environment using patient whole blood for pathogen detection and identification versus standard of care methods from blood culture.

The objective of this study is to determine the sensitivity and specificity of the Microbio InfectID-BSI qPCR kit by the evaluation of clinical blood samples versus standard of care methods from blood culture.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of neonates (less than 1 month of age), paediatrics (between 1 month and 17 years of age) or adults (≥18 years of age).
* Admitted to ICU, Emergency Department, or other medical wards for acute illness with medical decision to perform blood culture for suspicion of bloodstream Infection.
* Two additional EDTA blood sample/s collected from one anatomical site and at the same time as blood culture (two EDTA samples to be collected where possible).
* EDTA blood volume is ≥1mL.
* EDTA blood sample is stored according to Microbio's stability requirements.

Exclusion Criteria:

* No suspicion of blood stream infection (BSI).
* Any inclusion criterion not met.
* Multiple EDTA blood samples from the same patient.
* EDTA blood sample not obtained from the same anatomical site and at the same time as the blood culture sample.
* Subject has had an antimicrobial drug administered through the same port or central line as is used to collect the specimen.
* EDTA blood samples that have not been stored according to Microbio's sample stability requirements.
* EDTA blood volume <1mL.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study seeks to enroll neonates (less than 1 month of age), pediatrics (between 1 month and 17 years of age) and adults (>18 years of age) who are suspected to have a blood stream infection (BSI /Sepsis).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Determine the sensitivity and specificity of InfectID-BSI versus blood culture. | Through study completion, an average of 1 year
  The objective of this study is to determine the sensitivity and specificity of the Microbio InfectID-BSI qPCR kit by the evaluation of clinical blood samples versus standard of care methods from blood culture.
Determine the efficacy of detection and identification of the 26-pathogen panel in the InfectID-BSI assay versus standard of care blood culture. Using qPCR - a new molecular technology to identify the top 20 bacterial and 6 yeast sepsis causing species. | Through study completion, an average of 1 year
  The objective of the study is to determine the efficacy of the Microbio InfectID-BSI qPCR kit in a clinical laboratory environment using patient whole blood for pathogen detection and identification versus standard of care methods from blood culture. InfectID has it's own reporting software - InfectID-Client which is how the InfectID-BSI results will be reported for the study.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Indiana University Hospital, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - TriCore Reference Laboratories, Albuquerque, New Mexico
  - Vanderbilt University Medical Centre, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
- Australia (2):
  - The Prince Charles Hospital, Chermside, Queensland
  - The Princess Alexandra Hospital, Woolloongabba, Queensland
- Southwest Regional Laboratory, UK Health Security Agency, Bristol UK, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No